CLINICAL TRIAL: NCT03309943
Title: Neurobehavioral Substrates of Propranolol's Effects on Drug Cue Reactivity
Acronym: ProCue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00083809
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive propranolol (40 mg) or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Propranolol Capsule: 40 mg IR, administered 2x at separate laboratory sessions
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Placebo Capsule: No active ingredients, administered 2x at separate laboratory sessions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Participants will take one dose of Propranolol (40mg IR) on two separate occasions.
  Arms: Propranolol
Drug: Placebo — Participants will take one dose of Placebo on two separate occasions.
  Arms: Placebo

SUMMARY:
The central objective of this project is to obtain proof-of-concept data demonstrating the effects of propranolol (a beta-adrenergic antagonist) on neurobiological responses to personal smoking environments and behavioral responses in a laboratory smoking behavior task. Human cigarette smokers (N = 50) will take photographs of locations where they do and do not smoke cigarettes. They will then be randomly assigned to receive either propranolol (40 mg) or placebo prior to completing: A) An MRI session assessing neural responses to personal smoking/non-smoking environments, standard smoking/non-smoking environments and proximal smoking/non-smoking cues; and B) A laboratory session examining smoking behavior in response to environmental cues.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 55
* Generally healthy
* Right-handed
* Smoke >= 5 cigarettes/day of a brand delivering 0.5 mg nicotine (FTC method)
* Have been smoking regularly for >= 1 year, with a stable smoking pattern over the past 6 months
* Have an expired CO concentration of >= 10 ppm or urinary cotinine > 100 ng/ml
* Are able to identify at least 4 smoking and 4 non-smoking enviornments

Exclusion Criteria:

* Inability to attend all required sessions
* Significant health problems that would interfere with completion of study procedures
* Presence of conditions that would make MRI unsafe (e.g. pacemaker)
* Presence of exclusionary psychopathology based on MINI interview (current alcohol/substance use disorder moderate or severe pmild is allowable], any history of bipolar disorder or psychosis). Individuals in early remission from substance use disorder (not in a controlled environment) may also be allowed at the PIs discretion
* Current use of psychoactive medications per self-report or urine screen. Certain prescribed medications are allowable at the PI's discretion if appropriate documentation (e.g. copy of prescription or physician letter) is provided
* Positive breath alcohol concentraiton Pregnant, breastfeeding, or planning to become pregnant during the course of study
* Problems with vision that cannot be corrected with contacts or glasses
* Current regular use of smokeless tobacco, smoking cessation medications or non-combustible nicotine products (e.g. e-cigarettes)
* Plans to alter smoking pattern (e.g. reduction, uptake, cessation) during course of study
* Current use of beta-adrenergic medication
* Systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg (sitting or standing)
* Low resting heart rate (< 60 beats per minute)
* Abnormal EKG
* Presence of severe anemia (per complete blood count)
* Presence of electrolyte imbalance that could impact blood pressure (per metabolic panel)
* Presence of any other contraindications for propranolol (e.g. cardiovascular disease, bronchial asthma, prior allergic reaction)

Note that the above criteria reflect general guidelines for decision-making, but ultimate determinations are left to the discretion of the study physician. Presence of minor (e.g. asymptomatic bradycardia in the range of 50-60 in an otherwise healthy adult) or transient (e.g. electrolyte imbalance readily addressed via changes in fluid intake) may still be deemed eligible to participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Oliver, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Detailed protocols, datasets and additional information will be available from the Principal Investigator and research team upon request. In order to maintain compliance with HIPAA requirements (as well as university data security policies), all data will be de-identified according to HIPAA guidelines prior to being shared. Personal images themselves will not be made publicly available due to privacy concerns. However, a brief description of each image (e.g. "Front porch of home") will be made available. Data would be provided in widely accessible formats (e.g. csv/xls), along with a detailed data dictionary describing all elements and coding and study protocols.
Supporting Information: Study Protocol
Time Frame: We anticipate making data available within six months of study completion. It will be available for an indefinite period of time.
Access Criteria: Contact PI for details

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a laboratory setting at Duke University School of Medicine during a period ranging from January 2018 to June 2019.
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 22 | 22
Completed | 22 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Inappropriate behavior towards staff | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (9.6) | 35.0 (10.4) | 36.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 11 | 7 | 18
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes/day] — Self-reported average number of cigarettes smoked per day at screening (baseline) visit
  Cigarettes/day | 15.0 (6.1) | 15.4 (7.3) | 15.2 (6.6)
Fagerstrom Test for Cigarette Dependence [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Cigarette Dependence - This is an established self-report measure used to characterize the severity of nicotine dependence. Yes/no items are scored as 0 or 1 and multiple-choice items are scored from 0 to 3. These are summed to yield a total score ranging from 0 (no/minimal nicotine dependence) to 10 (severe nicotine dependence).
  units on a scale | 4.2 (1.7) | 5.4 (2.2) | 4.8 (2.0)
Contemplation Ladder (Motivation to Quit) [Mean (Standard Deviation); unit: units on a scale] — Contemplation Ladder - An established single-item measure of motivation to quit smoking. Participants rate themselves on a scale ranging from 0 (No thought of quitting) to 10 (Currently taking action to quit).
  units on a scale | 4.9 (2.5) | 3.3 (2.9) | 4.1 (2.8)
Number of Previous Quit Attempts [Mean (Standard Deviation); unit: quit-attempts] — Self-reported number of previous quit attempts based on a smoking history form collected at baseline (screening) visit.
  quit-attempts | 2.5 (2.3) | 2.0 (1.6) | 2.2 (2.0)
Education [Count of Participants; unit: Participants] — Self-reported educational attainment
  Participants
    Education <= High School Diploma | 10 | 8 | 18
    Education > High School Diploma | 12 | 12 | 24
Income [Count of Participants; unit: Participants] — Self-reported USUAL annual household income.
  Participants
    Usual Annual Income < $30,000 | 8 | 13 | 21
    Usual Annual income >= $30,000 | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: BOLD Activation to Smoking Cues - Amygdala
Description: BOLD activation in amygdala (% Signal Change). These are analyzed as separate units for each Trial Type (6 total: Proximal Non-Smoking, Proximal Smoking, Standard Environment Non-Smoking, Standard Environment Smoking, Personal Environment Non-Smoking, personal Environment Smoking), MRI Run (4 total: The task was divided into 4 runs to allow for participant breaks) and Brain Hemisphere (2 total: Left and Right). These are only presented by trial type as MRI Run and Brain Hemisphere are not variables of interest.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: Participants who completed the study. Excludes two additional participants in the placebo condition who had excessive motion artifact during scanning and could not be included in neuroimaging analyses.
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Units Other Than Participants: Trial Type, MRI Run, Brain Hemisphere
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
Number analyzed (Trial Type, MRI Run, Brain Hemisphere) | 1056 | 864
Percent Signal Change
  Non-Smoking Personal Environments | 0.002471 (0.367038) | 0.077325 (0.337887)
  Smoking Personal Environments | 0.009450 (0.384823) | 0.090345 (0.293101)
  Non-Smoking Standard Environments | 0.044903 (0.352711) | 0.042836 (0.341324)
  Smoking Standard Environments | 0.111746 (0.321235) | 0.161114 (0.355927)
  Non-Smoking Proximal | 0.066409 (0.386921) | 0.015171 (0.353829)
  Smoking Proximal | 0.025432 (0.378728) | 0.133363 (0.409809)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Mixed model analysis examining the effects of drug condition on response to smoking vs. non-smoking cues (collapsed across category - proximal, standard environment, personal environment). Data were analyzed using the underlying raw values versus collapsing them together; p = .019, Mixed Models Analysis; Adjusted for FTCD. Carried out using SPSS Mixed Models with a repeated statement and compound symmetry covariance structure

2. Primary Outcome: BOLD Activation to Smoking Cues - Anterior Insula
Description: BOLD activation in Anterior Insula (% Signal Change). These are analyzed as separate units for each Trial Type (6 total: Proximal Non-Smoking, Proximal Smoking, Standard Environment Non-Smoking, Standard Environment Smoking, Personal Environment Non-Smoking, personal Environment Smoking), MRI Run (4 total: The task was divided into 4 runs to allow for participant breaks) and Brain Hemisphere (2 total: Left and Right). These are only presented by trial type as MRI Run and Brain Hemisphere are not variables of interest.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Units Other Than Participants: Trial Type, MRI Run, Brain Hemisphere
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
Number analyzed (Trial Type, MRI Run, Brain Hemisphere) | 176 | 144
Percent Signal Change
  Non-Smoking Personal Environments | -0.179076 (0.288539) | -0.157851 (0.281748)
  Smoking Personal Environments | -0.127730 (0.293581) | -0.142636 (0.269551)
  Non-Smoking Standard Environments | -0.118271 (0.317144) | -0.152299 (0.326875)
  Smoking Standard Environments | -0.146114 (0.312662) | -0.149887 (0.282468)
  Non-Smoking Proximal | -0.085715 (0.331652) | -0.085873 (0.270967)
  Smoking Proximal | -0.086867 (0.352310) | -0.098181 (0.318646)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .830, Mixed Models Analysis; Adjusted for FTCD

3. Primary Outcome: BOLD Activation to Smoking Cues - Anterior Hippocampus
Description: BOLD activation in Anterior Hippocampus (% Signal Change). These are analyzed as separate units for each Trial Type (6 total: Proximal Non-Smoking, Proximal Smoking, Standard Environment Non-Smoking, Standard Environment Smoking, Personal Environment Non-Smoking, personal Environment Smoking), MRI Run (4 total: The task was divided into 4 runs to allow for participant breaks) and Brain Hemisphere (2 total: Left and Right). These are only presented by trial type as MRI Run and Brain Hemisphere are not variables of interest.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Units Other Than Participants: Trial Type, MRI Run, Brain Hemisphere
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
Number analyzed (Trial Type, MRI Run, Brain Hemisphere) | 176 | 144
Percent Signal Change
  Non-Smoking Personal Environments | 0.061001 (0.324934) | 0.095120 (0.271027)
  Smoking Personal Environments | 0.073925 (0.300800) | 0.088399 (0.267232)
  Non-Smoking Standard Environments | 0.133369 (0.315323) | 0.083638 (0.277520)
  Smoking Standard Environments | 0.171673 (0.289132) | 0.186590 (0.300916)
  Non-Smoking Proximal | 0.088852 (0.323655) | 0.000827 (0.280219)
  Smoking Proximal | 0.024626 (0.296327) | 0.095598 (0.291577)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .006, Mixed Models Analysis

4. Primary Outcome: BOLD Activation to Smoking Cues - Posterior Hippocampus
Description: BOLD activation in Posterior Hippocampus (% Signal Change). These are analyzed as separate units for each Trial Type (6 total: Proximal Non-Smoking, Proximal Smoking, Standard Environment Non-Smoking, Standard Environment Smoking, Personal Environment Non-Smoking, personal Environment Smoking), MRI Run (4 total: The task was divided into 4 runs to allow for participant breaks) and Brain Hemisphere (2 total: Left and Right). These are only presented by trial type as MRI Run and Brain Hemisphere are not variables of interest.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Units Other Than Participants: Trial Type, MRI Run, Brain Hemisphere
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
Number analyzed (Trial Type, MRI Run, Brain Hemisphere) | 176 | 144
Percent Signal Change
  Non-Smoking Personal Environments | 0.161077 (0.288481) | 0.185521 (0.262021)
  Smoking Personal Environments | 0.156684 (0.303924) | 0.166154 (0.252282)
  Non-Smoking Standard Environments | 0.137124 (0.304769) | 0.161655 (0.241679)
  Smoking Standard Environments | 0.179651 (0.256910) | 0.176196 (0.269538)
  Non-Smoking Proximal | 0.056247 (0.281092) | 0.053026 (0.271871)
  Smoking Proximal | 0.050077 (0.260461) | 0.121240 (0.262651)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .653, Mixed Models Analysis

5. Primary Outcome: BOLD Activation to Smoking Cues - Medial Prefrontal Cortex
Description: BOLD activation in Medial Prefrontal Cortex (% Signal Change). These are analyzed as separate units for each Trial Type (6 total: Proximal Non-Smoking, Proximal Smoking, Standard Environment Non-Smoking, Standard Environment Smoking, Personal Environment Non-Smoking, personal Environment Smoking), MRI Run (4 total: The task was divided into 4 runs to allow for participant breaks) and Brain Hemisphere (2 total: Left and Right). These are only presented by trial type as MRI Run and Brain Hemisphere are not variables of interest.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Units Other Than Participants: Trial Type, MRI Run, Brain Hemisphere
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
Number analyzed (Trial Type, MRI Run, Brain Hemisphere) | 176 | 144
Percent Signal Change
  Non-Smoking Personal Environments | 0.033030 (0.322540) | 0.012705 (0.409304)
  Smoking Personal Environments | 0.058184 (0.378236) | 0.060320 (0.313844)
  Non-Smoking Standard Environments | -0.078483 (0.350182) | -0.167025 (0.447513)
  Smoking Standard Environments | -0.068693 (0.311347) | -0.093598 (0.447743)
  Non-Smoking Proximal | -0.039529 (0.362686) | -0.109172 (0.422732)
  Smoking Proximal | -0.064034 (0.345958) | 0.015524 (0.413311)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .012, Mixed Models Analysis; Adjusted for FTCD

6. Primary Outcome: fMRI BOLD Connectivity
Description: Connectivity with right amygdala when viewing proximal smoking images, using a right anterior hippocampus seed region (psychophysiological interaction analysis; PPI). Larger values represent greater connectivity between these regions while viewing proximal smoking images.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PPI Index
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
PPI Index | -0.0740 (0.0769) | 0.0228 (0.0997)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Mixed model analysis examining the effects of drug condition on PPI indexes while viewing proximal smoking cues (which drove activation effects); p = .013, Mixed Models Analysis

7. Primary Outcome: Cue-Provoked Craving - Proximal Cues
Description: During MRI Scans, participants rated their craving in response to the question "While focusing on the place/object, I craved a cigarette." using a 1 (Do not agree) to 8 (Strongly agree) scale immediately following each image. Ratings were then averaged within each image category (total scale range of 1-8). Higher values represent greater craving.
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
units on a scale
  Non-Smoking | 2.866883 (1.566946) | 1.898148 (0.824614)
  Smoking | 6.103084 (1.618450) | 6.547619 (1.685597)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Repeated Measures ANCOVA analysis examining condition differences (adjusting for FTCD score); p = .024, Repeated Measures ANCOVA; Adjusted for FTCD

8. Primary Outcome: Cue-Provoked Craving - Standard Environment Images
Description: as for outcome 7
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 18
units on a scale
  Non-Smoking | 2.673052 (1.681618) | 1.763889 (0.644389)
  Smoking | 4.666937 (1.588874) | 4.868056 (1.716846)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Repeated Measures ANCOVA analysis examining condition differences (adjusting for FTCD score); p = .086, Repeated Measures ANCOVA; Adjusted for FTCD score

9. Primary Outcome: Cue-Provoked Craving - Personal Environment Cues
Description: as for outcome 7
Time Frame: MRI Scan: 2-3 hours post-administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 20
units on a scale
  Non-Smoking | 3.369318 (1.802147) | 2.965278 (1.668703)
  Smoking | 6.045996 (1.457661) | 6.638889 (1.569405)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Repeated Measures ANCOVA analysis examining condition differences (adjusting for FTCD score); p = .140, Repeated Measures ANCOVA; Adjusted for FTCD score

10. Secondary Outcome: Laboratory Visit - Self-Reported Craving
Description: Self-reported craving to smoke following presentation of personal smoking environments (prior to ad-lib smoking period). Assessed using the average rating across four questions drawn from the Questionnaire on Smoking Urges: (1) While focusing on those places...nothing would have been better than smoking a cigarette; (2) While focusing on those places...I had the urge for a cigarette; (3) While focusing on those places...all I wanted right then was a cigarette; (4) While focusing on those places...I craved a cigarette. Participants rated each item on an 11-point scale ranging from 0 (Do not agree) to 100 (Strongly agree) in 10-point intervals. These ratings were averaged across items for analysis. higher values represent greater craving.
  Tiffany, S. T., & Drobes, D. J. (1991). The development and initial validation of a questionnaire on smoking urges. British Journal of addiction, 86(11), 1467-1476.
Time Frame: Lab Task: 2-3 hours post-administration
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 20
units on a scale | 7.3 (2.7) | 7.9 (3.0)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Standard ANCOVA analysis examining condition differences (adjusting for baseline craving and FTCD score); p = .556, ANCOVA; Adjusted for baseline craving and FTCD score

11. Secondary Outcome: Laboratory Visit - # Cigarette Puffs
Description: Number of cigarette puffs taken during ad lib smoking period while participants view images of their personal smoking environment. Smoking was video recorded and puffs were coded by two raters.
Time Frame: Lab Task: 2-3 hours post-administration
Population: Participants who completed the study. Data from one participant in the placebo condition was lost due to technical problems with the recording.
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 19
Puffs | 15.2 (7.1) | 17.7 (9.8)
Statistical Analysis 1: Comparison: Propranolol vs Placebo; Test type: Superiority — Standard ANCOVA analysis examining condition differences (adjusting for FTCD score); p = .463, ANCOVA — Adjusted for FTCD score only

ADVERSE EVENTS:
Time Frame: This is an acute administration study with an approved medication with a well-established safety profile. Adverse events were assessed over the 1-3 month period in which participants were engaged in the project, primarily for purposes of ensuring new contraindications did not emerge prior to drug administration vs concerns about adverse events related to the drug itself.
Description: Participants abstain from smoking for 24 hours before the MRI visit and 6 hours before the laboratory visit. Symptoms of nicotine withdrawal are assessed but are not considered adverse events. Participant self-report of any newly-onset or worsening medical problems during their time of participation are considered adverse events. Repeat blood draws were occasionally necessary but are also not considered adverse events.
Arm/Group | Propranolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=22) | Placebo (N=22)
Dog Bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported having been bitten by a dog prior to their MRI visit.
Wrist Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant arrived to MRI appointment in a wrist brace and reported they had sprained their wrist two days prior to the appointment.

LIMITATIONS AND CAVEATS:
This was a pilot study with a small sample size. A between-subjects design was used with no baseline scan for comparison. No clinical endpoints were examined - results are limited to neuroimaging and behavioral task outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03309943/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT03309943/Prot_SAP_001.pdf